CLINICAL TRIAL: NCT03716427
Title: A Fixed-Sequence Trial to Examine the Effect of Multiple-Dose CT1812 Administration on Standard Probes of CYP2C19 (Omeprazole), CYP2C9 (Tolbutamide), CYP2D6 (Dextromethorphan), and CYP3A4/5 (Midazolam) Activity in Healthy Adult Volunteers
Brief Title: Drug Interaction Study of CT1812 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COG0103
Record Dates: First submitted 2018-08-16; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Tolbutamide; Dextromethorphan; Omeprazole; Midazolam

STUDY DESIGN:
Intervention Model Description: This is Phase 1, single-center, open-label, single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of 4 probe drugs (tolbutamide, midazolam, dextromethorphan and omeprazole)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Treatment- CT1812 560 mg (Experimental): Single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of 4 probe drugs (tolbutamide, midazolam, dextromethorphan and omeprazole)
  Interventions: Drug: CT1812; Drug: tolbutamide; Drug: dextromethorphan; Drug: Omeprazole; Drug: midazolam

INTERVENTIONS:
Drug: CT1812
Drug: tolbutamide — Single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of tolbutamide
Drug: dextromethorphan — Single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of dextromethorphan
Drug: Omeprazole — Single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of omeprazole
Drug: midazolam — Single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of midazolam

SUMMARY:
This is Phase 1, single-center, open-label, single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of 4 probe drugs (tolbutamide, midazolam, dextromethorphan and omeprazole).

DETAILED DESCRIPTION:
This is Phase 1, single-center, open-label, single-sequence drug-drug interaction study to determine the effect of CT1812 (560 mg) once daily on the pharmacokinetics of 4 probe drugs (tolbutamide, midazolam, dextromethorphan and omeprazole).

Each subject will qualify for entry into the study within 35 days before admission to the clinical unit. Subjects will check into the clinical unit on Day -3 for baseline assessments. Each subject will receive a single dose of each of the probe drugs on Day -2 as a 'cocktail'. A single dose of CT1812 and each of the probe drugs will be co-administered on Day 6. On Days 1 through 5, subjects will receive a single daily dose of CT1812.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to initiation of any study-related procedures.
2. Men and women ≥ 18 and ≤ 55 years of age
3. In good health as determined by medical history, physical exam, laboratory examinations, ECG, and vital signs
4. BMI between 18 and 35 kg/m2, inclusive
5. Have a normal 12-lead electrocardiogram, without any clinically significant abnormalities of rate, rhythm or conduction
6. Non-smokers; defined as not having smoked in the previous 6 months
7. Women who are neither pregnant (negative pregnancy test) nor nursing, and are either:

   1. Surgically sterile (bilateral tubal ligation, hysterectomy), or
   2. Postmenopausal with last natural menses greater than 12 months, or
   3. Premenopausal and using an acceptable barrier form of birth control from screening until two-weeks post discharge. Acceptable forms of birth control include abstinence and any double combination of: hormonal contraceptive, intrauterine device (IUD), male or female condom, diaphragm, sponge, and cervical cap. Spermicides may be used, but is not considered one of the required double barrier methods. All premenopausal female subjects (regardless of whether they are surgically sterile) must have a negative serum pregnancy test at screening and baseline.

Exclusion Criteria:

1. Known hypersensitivity or allergy to omeprazole, tolbutamide, dextromethorphan, midazolam, or CT1812
2. Absence of one functional allele for CYP2D6, CYP2C9 or CYP2C19 at screening
3. Any disease or condition (medical or surgical) which, in the opinion of the Investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
4. The presence of abnormal laboratory values which are considered clinically significant
5. Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2)
6. Received an investigational drug within a period of 30 days prior to enrollment in the study
7. Received any drug therapy within 2 weeks prior to administration of the first dose of any study-related treatment. This exclusion is extended to 4 weeks for any drugs known to induce or inhibit hepatic drug metabolism.
8. Consumption of alcohol within 14 days prior to dose administration or during any in-patient period
9. A positive urine drug screen including ethanol, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and opiates
10. Any history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid within the past two years, or any history of drug abuse or addiction within the past two years
11. A history of difficulty with donating blood
12. Donated whole blood within 45 days or blood products within 7 days prior to enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Area under the plasma-concentration time curve of CT1812 (Day 6) compared to the baseline values (Day -2) | 10 days
  Single dose (Day -2 and Day 6) pharmacokinetic parameter Area under the plasma-concentration time curve

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Galley, Study Director — Cognition Therapeutics, Inc.
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No